CLINICAL TRIAL: NCT02198378
Title: Analgesia of Acute Coronary Syndromes With ST-segment Elevation in a Pre-hospital Setting. Randomized Non-inferiority Trial of the Association MEOPA + Paracetamol Versus Morphine.
Brief Title: Comparison of MEOPA + Paracetamol Versus Morphine Treatment in Acute Coronary Syndrome Analgesia.
Acronym: SCADOLII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/13/7050; 13705001 (Other Grant/Funding Number: French Ministry of Health, PHRC 2013)
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome
Keywords: premixed nitrous oxide and oxygen; pain; prehospital setting; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Pain | interventions — Meopa; Acetaminophen; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Morphine group: administration of morphine will start with a 0.05 mg/kg bolus followed by reinjection of 2 mg every 5 minutes until effective analgesia is obtained, defined as NRS ≤ 3.
  Interventions: Drug: Morphine
- MEOPA and paracetamol (Experimental): The patient will be equipped with a facemask delivering MEOPA.The gas flow received by the patient is adapted to his/her ventilation.
  During the same time, an intravenous injection of 1 g paracetamol will be administered.
  Interventions: Drug: MEOPA and paracetamol

INTERVENTIONS:
Drug: MEOPA and paracetamol — The patient will be equipped with a facemask after he/she has been informed. The facemask is adapted to the patient. The patient breathes normally in the mask which is held in place by a member of the SMUR team who has received previous training in use of MEOPA. The gas flow received by the patient is adapted to his/her ventilation.
  Other Names: Entonox 170 bar
  Arms: MEOPA and paracetamol
Drug: Morphine — Bolus of 2 mg intravenously if EN = 4 or 5 and 3 mg bolus if EN> 6 followed by reinjection of 2mg every 5 minutes until effective analgesia.
  Other Names: Morphine Renaudin 1mg/ml
  Arms: Morphine

SUMMARY:
In the management of acute coronary syndromes with ST-segment elevation (STEMI), early analgesia reduces the effects of hyperadrenalism which increases the size of myocardial infarction. In order to reduce pain intensity, the recommendations advocate emergency use of morphine. In STEMI patients, other analgesic treatments could provide analgesia that is at least as effective as morphine. The equimolar oxygen/nitrous oxide mixture (MEOPA) is widely used in emergency medicine and has minor secondary effects that are very rapidly reversible when inhalation is discontinued. Used in association with paracetamol, it could be an at least equally effective alternative to the use of morphine.

DETAILED DESCRIPTION:
The investigators wish to compare the use of morphine according to current recommendations with the use of MEOPA associated with intravenous paracetamol in the management of patients with STEMI. The investigators hypothesize that the association of MEOPA and paracetamol, which is easy to use in a pre-hospital setting, will give patients pain relief as effectively as morphine.

This alternative treatment would avoid the use of morphine, whose potentially damaging consequences on myocardial function have been suggested by experimental studies and by an observational study. The physician of the mobile emergency team (SMUR) verifies the inclusion and non- inclusion criteria for the study. The patient must present STEMI defined in accordance with the recommendations and chest pain of intensity ≥ 4 on the NRS. The specific treatment for STEMI will be given before inclusion in the study, with the exception of analgesic treatment. In particular, inclusion in the study must not delay the initiation of strategies of recanalization and reperfusion.

The SMUR physician in charge of the patient will administer the treatment defined by randomization.

After 30 minutes, the patient will be managed in accordance with the recommendations and will be hospitalized, generally in a cardiology intensive care unit. At one month, the clinical research technician will record the patient's vital status and collect the patient's hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Patient with STEMI < 12 h treated before hospital admission and pain ≥ 4 on the numerical rating scale.

Exclusion Criteria:

* Acute severe hemodynamic, respiratory or neurological failure
* Heart failure: Killip class III and IV
* Known allergy to morphine or nitrous oxide
* Patient who has already received morphine or MEOPA before the arrival of the hospital team during the 4 hours preceding the pre-hospital intervention
* Contraindications to nitrous oxide
* Patient unable to assess pain intensity on the numerical rating scale
* Patient under legal guardianship
* Pregnancy
* Patient transported by air ambulance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Effective analgesia (NRS score≤ 3) at 30 minutes after the start of analgesia | 30 minutes after randomisation.
  The primary outcome measure is effective analgesia, defined by the consensus conference as an NRS score ≤ 3 at 30 minutes after the start of analgesia.

SECONDARY OUTCOMES:
Adverse event | all 5 minutes during 30 minutes
  Occurrence of an adverse effect, in particular, respiratory depression (RR, respiratory rate < 10 cycles par minute or respiratory score ≥ R1), nausea, vomiting, sedation (sedation scale (EDS) score ≥2), dizziness, pruritus.
NRS distribution | 30 minutes after randomization
  Distribution of the NRS at 30 minutes and on arrival at the cardiology unit
Effective analgesia | all 5 minutes during 30 minutes
  The time of effective analgesia will be defined for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Charpentier, PH,MD, Principal Investigator — University Hospital, Toulouse
Locations (40):
- France (39):
  - Centre Hospitalier d'Agen, Agen
  - Centre Hospitalier Jean Minjoz, Besançon
  - CHU Avicenne, Bobigny
  - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Bourg-en-Bresse, Bourg-en-Bresse
  - Centre Hospitalier de Chambéry, Chambéry
  - Centre Hospitalier Louis Pasteur, Chartres
  - Centre Hospitalier Chateauroux, Châteauroux
  - CHU d'Estaing, Clermont-Ferrand
  - Centre Hospitalier Beaujon, Clichy
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Dijon, Dijon
  - Centre Hospitalier du Val d'Ariège, Foix
  - Centre Hospitalier Raymond Poincaré, Garches
  - Centre Hospitalier de Grenoble, Grenoble
  - Centre Hospitalier Départemental La Roche/Yon, La Roche-sur-Yon
  - CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Centre Hospitalier Edouard Herriot, Lyon
  - Centre Hospitalier de la Timone, Marseille
  - Centre Hospitalier Marc Jacquet, Melun
  - CHR Bon Secours, Metz
  - CHRU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Centre Hospitalier de Nice, Nice
  - Centre Hospitalier Necker, Paris
  - Centre Hospitalier Pitié-Salpétrière, Paris
  - Groupe hospitamier Lariboisière-Fernand Widal-St-Louis, Paris
  - CHU Poitiers, Poitiers
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier Annecy-Gennevois, Pringy
  - Centre Hospitalier Comminges Pyrénées, Saint-Gaudens
  - Centre Hospitalier Poulon la Seyne-sur-mer, Toulon
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours
  - Centre Hospitalier de Valence, Valence
  - Centre Hospitalier Lucien Hussel, Vienne
- CHU Félix Guyon, Saint-Denis, Reunion

REFERENCES:
- [Background] Danchin N, Puymirat E, Aissaoui N, Adavane S, Durand E. [Epidemiology of acute coronary syndromes in France and in Europe]. Ann Cardiol Angeiol (Paris). 2010 Dec;59 Suppl 2:S37-41. doi: 10.1016/S0003-3928(10)70008-1. French. PMID 21237321
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764
- [Background] Task Force for Diagnosis and Treatment of Non-ST-Segment Elevation Acute Coronary Syndromes of European Society of Cardiology; Bassand JP, Hamm CW, Ardissino D, Boersma E, Budaj A, Fernandez-Aviles F, Fox KA, Hasdai D, Ohman EM, Wallentin L, Wijns W. Guidelines for the diagnosis and treatment of non-ST-segment elevation acute coronary syndromes. Eur Heart J. 2007 Jul;28(13):1598-660. doi: 10.1093/eurheartj/ehm161. Epub 2007 Jun 14. No abstract available. PMID 17569677
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Canadian Cardiovascular Society; American Academy of Family Physicians; American College of Cardiology; American Heart Association; Antman EM, Hand M, Armstrong PW, Bates ER, Green LA, Halasyamani LK, Hochman JS, Krumholz HM, Lamas GA, Mullany CJ, Pearle DL, Sloan MA, Smith SC Jr, Anbe DT, Kushner FG, Ornato JP, Pearle DL, Sloan MA, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA 2004 guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):210-47. doi: 10.1016/j.jacc.2007.10.001. No abstract available. PMID 18191746
- [Derived] Charpentier S, Galinski M, Bounes V, Ricard-Hibon A, El-Khoury C, Elbaz M, Ageron FX, Manzo-Silberman S, Soulat L, Lapostolle F, Gerard A, Bregeaud D, Bongard V, Bonnefoy-Cudraz E; SCADOL II investigators. Nitrous oxide/oxygen plus acetaminophen versus morphine in ST elevation myocardial infarction: open-label, cluster-randomized, non-inferiority study. Scand J Trauma Resusc Emerg Med. 2020 May 12;28(1):36. doi: 10.1186/s13049-020-00731-y. PMID 32398160